CLINICAL TRIAL: NCT02075099
Title: Evaluation of the Efficiency of a Hydration by Isotonic Solution With or Without Muscular Exercise of the Fainting Whole Blood Donors
Brief Title: Evaluation of the Efficiency of Hydration by Isotonic Solution in the Prevent of the Fainting Whole Blood Donors
Acronym: EVASION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Etablissement Français du Sang (Other)
Collaborators: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: DCIC 13 53
Record Dates: First submitted 2014-02-14; First posted 2014-03-03 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-02

CONDITIONS: Fainting; Presyncope; Syncopal Episode
Keywords: whole blood donation; donation water drink; isotonic drink; presyncopal and syncopal reactions
MeSH Terms: conditions — Syncope

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Isotonic drink (Experimental): Predonation hydratation with 500 ml of isotonic drink, to drinking in immediate predonation.
  (The half of included donors will do "tensing exercises" during the blood whole donation and the other half will do "no tensing exercises")
  Interventions: Other: tensing exercises; Other: No tensing exercises
- mineral water (Experimental): Predonation hydratation with 500 ml of mineral water to drinking in immediate predonation whole blood.
  (The half of included donors will do "tensing exercises" during the blood whole donation and the other half will do "no tensing exercises")
  Interventions: Other: tensing exercises; Other: No tensing exercises
- Advices (Active Comparator): Advices of drinking water or fruit juice glass(es) in immediate predonation whole blood.
  (The half of included donors will do "tensing exercises" during the blood whole donation and the other half will do "no tensing exercises")
  Interventions: Other: tensing exercises; Other: No tensing exercises

INTERVENTIONS:
Other: tensing exercises — Donors will do tensing exercises during blood donation
Other: No tensing exercises — Donors will not do tensing exercises during blood donation - control arm

SUMMARY:
Blood donation is a generous act carried out by healthy male and female volunteer donors. The safety of blood donation in France is based on rigorous well documented biological and medical criteria, in particular concerning the volume of blood to be taken. While whole blood donation is very safe, some donors experience faintness during or after donation. Any injury resulting from a fall increases its seriousness, especially when it happens outside the donation site.

According to various studies, adverse reactions are experienced by between 0.28% and 2.72% of all donors and occur in all categories (sex and age).

A retrospective evaluation of the frequency of faintness incidents on during whole blood donation over 2012 in the Rhone Alpes' region of France shows a frequency ranging from 1.05% in mobile donation units in towns to 4.24% in donation units in high schools, with no reporting of delayed incidents of faintness by this donor population.

DETAILED DESCRIPTION:
Despite precautions including advice to donors to drink some water before blood donation, fainting events still occur. They can have an impact on the frequency of donation as well as on the blood donor's motivation and that in their close entourage. This impact should not be overlooked in the context of the increasing need for blood components and tighter budgets..

In some other national health systems, the donor is given a drink shortly before giving blood and / or donors are advised to do lower-body muscle tensing exercises whilst giving blood.

The present study has a factorial design and compares 3 arms for hydration criteria and 2 arms for exercise criteria with cluster randomization (1 cluster = 1 blood donation unit). The randomization plan will be stratified according to the type of EFS donation unit (French Blood Donation service: Etablissement Français du Sang): Fixed/Mobile unit; and also on the location of the of mobile blood donation unit: in companies, towns or schools. In the latter, the blood donors have a potentially higher risk of presyncopal or syncopal reactions.

3 arms:

* 500mL of an isotonic drink to be drunk immediately before blood donation
* 500mL of slightly mineralized water to be drunk immediately before blood donation
* Advice to drink one glass of fruit juice or water before blood donation In the 3 arms, the centralized randomization will balance the numbers of blood donations in which the donors will perform lower-body muscle tensing exercises , or not, during the blood donation.

Main objective:

To assess the impact of preventive measures, including rapid hydration with 500mL of an isotonic drink versus hydration with 500mL of water or simple advice to have a drink; and advice to perform lower-body muscle tensing exercises during the whole blood donation, on the prevention of presyncopal and syncopal reactions during blood donation and in the following 48 hours.

ELIGIBILITY:
Inclusion Criteria:

- Whole blood donors , in fixed site or mobile collection

* 18-year-old and less than 71 years
* Donor with weight > in 50 kg and height> 135 cms
* Whole Blood donors having had an interview with a doctor of the EFS and declared capable
* Donors for phone contact in 7 days following the donation

Exclusion Criteria:

* Collection by an autonomous mobile blood collection unit (with independent management and sample storage)
* Donor with an immobilization, even partial, of a lower limb.
* Donor allergic to shellfish, gluten, milk or soya.
* Donor under judicial protection or other administrative control.

Ages: 18 Years to 71 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4825 (Actual)
Dates: Start 2014-01; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Accumulated incidence of presyncopal and syncopal reactions during blood donation, while still at the blood donation whole and within 48 hours of the blood donation, that required the donor to be placed in a 'Trendelenburg' position | At the time of inclusion and at 48 hours after the blood donation
  Symptoms of presyncopal reactions (blurring of vision, insensitivity to ambient noises, generalized weakness, paleness, nausea) and syncopal reactions that required the donor to be placed in the 'Trendelenburg' position
  * Presyncopal and syncopal symptoms requiring interruption of the blood donation
  * Vomiting
  * Unconsciousness with interruption of blood donation, with no other consequences and no specific treatment.
  * Convulsions
  * Leak of urine
  * Unconsciousness with interruption of blood donation with no other consequences, but with medical treatment by an oral route.
  * Unconsciousness with interruption of blood donation with no other consequences, but requiring a perfusion or intravenous treatment.
  * Unconsciousness immediately post donation with or without consequences
  * Presyncopal and syncopal reactions with or without consequences within the 48 hours after the blood donation
  * Angina, infarct
  * Death

SECONDARY OUTCOMES:
daily activities | 48 hours after the blood donation
  Evaluation of the impact of whole blood donation assess by :
  Modification of daily habits. Fatigue assessment scale for healthy subjects. Unusual fatigue depending on the type of proposed prevention (drinks and exercises).
presyncopal and syncopal reactions of all donors | inclusion and 48 hours after the blood donation
  This concerns presyncopal and syncopal reactions that required the donor to lie down in the Trendelenburg position and any further intervention.
  We will compare the occurrence of presyncopal and syncopal reactions during the blood donation, or immediately post-donation, while still in the blood donation center, and within 48 hours following blood donation.
  We will analysed separate from that of the main criterion in three periods: during the donation, immediate post donation, late post donation.
presyncopal and syncopal reactions in the population of young donors (in schools) | 48 hours after the blood donation
  Main criteria analyzed in the sub-population of blood donation at schools Evaluate the rate of presyncopal and syncopal reactions after the donation, but within 48 hours, in the population of young donors attending blood collection centers in schools.
presyncopal or syncopal reactions influence on subsequent blood donation | year which follows the blood donation
  Evaluate the influence of the occurrence of presyncopal or syncopal reactions on subsequent blood donation or not.
  Renewal of blood donation within one year (from the EFS database)
Recurrence of presyncopal or syncopal reactions | year which follows the blood donation
  Presyncopal and syncopal reactions during a following blood donation made within one year and listed in the EFS donor safety database Evaluate whether the occurrence of presyncopal or syncopal reactions is a predictor of recurrence during the next blood donation
Explanatory variables of presyncopal and syncopal reactions | 7 days after last donor inclusion
  Variables linked to the presyncopal and syncopal reactions as defined by the main criterion Explanatory variables: the characteristics of the donor (age, sex, number of previous blood donations), the circumstances of the blood donation (work or effort before the blood donation, the time of day of the blood donation, the quality of the post donation snack (sweet/salty) etc. and the characteristics of the blood donation unit/center (fixed/mobile, school/company/town, room/ mobile blood donation unit, size of the town, place of blood donation.
subgroup analysis on collection unit characteristics | 7 days after last donor inclusion
  subgroup analyses of the primary and secondary endpoints according to the characteristics of the collection unit used in the stratification of randomization of donors.
medium term impact of the donation | 7 days after the blood donation
  Main criterion and secondary criteria assessed at day 7 by phone call to the donor
Restless legs syndrome | months before the blood donation
  during phone call to the donor at day 7, questions will be asked about possible or probable RLS (Restless Legs Syndrome). Classification of Bryan R. Spencer (Transfusion August 2013) will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Chrystelle Morand, MD, Principal Investigator — EFS Rhone Alpes - Site Grenoble; Nicole Coudurier, MD, Principal Investigator — EFS LYON; Marie-Claude Bourboul, MD, Principal Investigator — EFS Rhone Alpes- Site Lyon; Debost Michèle, MD, Principal Investigator — EFS Rhone Alpes-site Lyon; Isabelle Michaud-Bauda, MD, Principal Investigator — EFS Rhone Alpes- site Grenoble
Locations (2):
- France (2):
  - EFS Grenoble, Grenoble
  - EFS Lyon, Lyon

REFERENCES:
- [Background] V. Candas, B. Bothorel : Hydratation, travail et chaleur. , INRS CDU 613-3 Fiche d'hygiène de vie au travail, Cahier de notes documentaires n° 135, 2ème trimestre 1989 : 241 - 245
- [Background] France CR, France JL, Kowalsky JM, Ellis GD, Copley DM, Geneser A, Frame-Brown T, Venable G, Graham D, Shipley P, Menitove JE. Assessment of donor fear enhances prediction of presyncopal symptoms among volunteer blood donors. Transfusion. 2012 Feb;52(2):375-80. doi: 10.1111/j.1537-2995.2011.03294.x. Epub 2011 Aug 16. PMID 21848969
- [Background] Eder AF, Hillyer CD, Dy BA, Notari EP 4th, Benjamin RJ. Adverse reactions to allogeneic whole blood donation by 16- and 17-year-olds. JAMA. 2008 May 21;299(19):2279-86. doi: 10.1001/jama.299.19.2279. PMID 18492969
- [Background] P. Tomasulo, M. Bravo et H. Kamel : Time course of vasovagal syncope with whole blood donation. ISBT Science Series, 2010 ; 5 : 52 - 58
- [Background] Wieling W, France CR, van Dijk N, Kamel H, Thijs RD, Tomasulo P. Physiologic strategies to prevent fainting responses during or after whole blood donation. Transfusion. 2011 Dec;51(12):2727-38. doi: 10.1111/j.1537-2995.2011.03202.x. Epub 2011 Jun 3. PMID 21645008
- [Background] Kowalsky JM, France JL, Wissel ME, France CR. Effect of applied muscle tension on cerebral oxygenation in female blood donors. Transfusion. 2011 Aug;51(8):1802-8. doi: 10.1111/j.1537-2995.2011.03075.x. Epub 2011 Mar 7. PMID 21382044
- [Background] Eder AF. Improving safety for young blood donors. Transfus Med Rev. 2012 Jan;26(1):14-26. doi: 10.1016/j.tmrv.2011.07.008. Epub 2011 Aug 26. PMID 21872427
- [Background] Eder AF. Current efforts to reduce the risk of syncope among young blood donors. Curr Opin Hematol. 2012 Nov;19(6):480-5. doi: 10.1097/MOH.0b013e328358b15c. PMID 22954724
- [Background] van den Berg K, Lam J, Bruhn R, Custer B, Murphy EL. Water administration and the risk of syncope and presyncope during blood donation: a randomized clinical trial. Transfusion. 2012 Dec;52(12):2577-84. doi: 10.1111/j.1537-2995.2012.03631.x. Epub 2012 Apr 4. PMID 22486209
- [Background] Physiologie Humaine 3e édition Hervé Guénard, ed Pradel. Rein : 307 - 313
- [Background] Eder AF, Notari EP 4th, Dodd RY. Do reactions after whole blood donation predict syncope on return donation? Transfusion. 2012 Dec;52(12):2570-6. doi: 10.1111/j.1537-2995.2012.03666.x. Epub 2012 Apr 27. PMID 22536827
- [Background] Eder A. Evidence-based selection criteria to protect blood donors. J Clin Apher. 2010;25(6):331-7. doi: 10.1002/jca.20257. Epub 2010 Sep 7. PMID 20824625
- [Background] Eder AF, Dy BA, Kennedy JM, Notari Iv EP, Strupp A, Wissel ME, Reddy R, Gibble J, Haimowitz MD, Newman BH, Chambers LA, Hillyer CD, Benjamin RJ. The American Red Cross donor hemovigilance program: complications of blood donation reported in 2006. Transfusion. 2008 Sep;48(9):1809-19. doi: 10.1111/j.1537-2995.2008.01811.x. Epub 2008 Jul 9. PMID 18631167
- [Background] Bravo M, Kamel H, Custer B, Tomasulo P. Factors associated with fainting: before, during and after whole blood donation. Vox Sang. 2011 Nov;101(4):303-12. doi: 10.1111/j.1423-0410.2011.01494.x. Epub 2011 May 3. PMID 21535440
- [Background] Carneiro-Proietti AB, Sabino EC, Sampaio D, Proietti FA, Goncalez TT, Oliveira CD, Ferreira JE, Liu J, Custer B, Schreiber GB, Murphy EL, Busch MP. Demographic profile of blood donors at three major Brazilian blood centers: results from the International REDS-II study, 2007 to 2008. Transfusion. 2010 Apr;50(4):918-25. doi: 10.1111/j.1537-2995.2009.02529.x. Epub 2009 Dec 10. PMID 20003051
- [Background] Trouern-Trend JJ, Cable RG, Badon SJ, Newman BH, Popovsky MA. A case-controlled multicenter study of vasovagal reactions in blood donors: influence of sex, age, donation status, weight, blood pressure, and pulse. Transfusion. 1999 Mar;39(3):316-20. doi: 10.1046/j.1537-2995.1999.39399219291.x. PMID 10204597
- [Background] Wiltbank TB, Giordano GF, Kamel H, Tomasulo P, Custer B. Faint and prefaint reactions in whole-blood donors: an analysis of predonation measurements and their predictive value. Transfusion. 2008 Sep;48(9):1799-808. doi: 10.1111/j.1537-2995.2008.01745.x. Epub 2008 May 14. PMID 18482188
- [Background] Eder AF, Dy BA, Kennedy JM, Perez J, Demaris P, Procaccio A, Benjamin RJ. Improved safety for young whole blood donors with new selection criteria for total estimated blood volume. Transfusion. 2011 Jul;51(7):1522-31. doi: 10.1111/j.1537-2995.2011.03143.x. Epub 2011 Apr 29. PMID 21534981
- [Background] Newman B, Tommolino E, Andreozzi C, Joychan S, Pocedic J, Heringhausen J. The effect of a 473-mL (16-oz) water drink on vasovagal donor reaction rates in high-school students. Transfusion. 2007 Aug;47(8):1524-33. doi: 10.1111/j.1537-2995.2007.01293.x. PMID 17655598
- [Background] Ando S, Kawamura N, Matsumoto M, Dan E, Takeshita A, Murakami K, Kashiwagi S, Kiyokawa H. Simple standing test predicts and water ingestion prevents vasovagal reaction in the high-risk blood donors. Transfusion. 2009 Aug;49(8):1630-6. doi: 10.1111/j.1537-2995.2009.02189.x. PMID 19413739
- [Background] France CR, Ditto B, Wissel ME, France JL, Dickert T, Rader A, Sinclair K, McGlone S, Trost Z, Matson E. Predonation hydration and applied muscle tension combine to reduce presyncopal reactions to blood donation. Transfusion. 2010 Jun;50(6):1257-64. doi: 10.1111/j.1537-2995.2009.02574.x. Epub 2010 Jan 22. PMID 20113455
- [Background] Tomasulo P, Kamel H, Bravo M, James RC, Custer B. Interventions to reduce the vasovagal reaction rate in young whole blood donors. Transfusion. 2011 Jul;51(7):1511-21. doi: 10.1111/j.1537-2995.2011.03074.x. Epub 2011 Mar 7. PMID 21382043
- [Background] Scott EM, Greenwood JP, Stoker JB, Gilbey SG, Mary DA. Water drinking and sympathetic activation. Lancet. 2000 Dec 9;356(9246):2013. doi: 10.1016/S0140-6736(05)72987-1. No abstract available. PMID 11130550
- [Background] A. F. Eder : can we improve safety for young blood donors ?. ISBT Science Series 2012;7:226-229
- [Background] Custer B, Rios JA, Schlumpf K, Kakaiya RM, Gottschall JL, Wright DJ; NHLBI Retrovirus Epidemiology Donor Study-II (REDS-II). Adverse reactions and other factors that impact subsequent blood donation visits. Transfusion. 2012 Jan;52(1):118-26. doi: 10.1111/j.1537-2995.2011.03216.x. Epub 2011 Jun 17. PMID 21682732
- [Background] France CR, France JL, Wissel ME, Ditto B, Dickert T, Himawan LK. Donor anxiety, needle pain, and syncopal reactions combine to determine retention: a path analysis of two-year donor return data. Transfusion. 2013 Sep;53(9):1992-2000. doi: 10.1111/trf.12069. Epub 2013 Jan 11. PMID 23305267
- [Background] France CR, France JL, Himawan LK, Stephens KY, Frame-Brown TA, Venable GA, Menitove JE. How afraid are you of having blood drawn from your arm? A simple fear question predicts vasovagal reactions without causing them among high school donors. Transfusion. 2013 Feb;53(2):315-21. doi: 10.1111/j.1537-2995.2012.03726.x. Epub 2012 Jun 7. PMID 22670781
- [Background] Veldhuizen I, Atsma F, van Dongen A, de Kort W. Adverse reactions, psychological factors, and their effect on donor retention in men and women. Transfusion. 2012 Sep;52(9):1871-9. doi: 10.1111/j.1537-2995.2011.03551.x. Epub 2012 Feb 10. PMID 22321030
- [Background] Ditto B, France CR, Albert M, Byrne N, Smyth-Laporte J. Effects of applied muscle tension on the likelihood of blood donor return. Transfusion. 2009 May;49(5):858-62. doi: 10.1111/j.1537-2995.2008.02067.x. Epub 2009 Jan 21. PMID 19175551
- [Background] Kamel H, Tomasulo P, Bravo M, Wiltbank T, Cusick R, James RC, Custer B. Delayed adverse reactions to blood donation. Transfusion. 2010 Mar;50(3):556-65. doi: 10.1111/j.1537-2995.2009.02397.x. Epub 2009 Oct 5. PMID 19804573
- [Background] Ditto B, France CR, Holly C. Applied tension may help retain donors who are ambivalent about needles. Vox Sang. 2010 Apr;98(3 Pt 1):e225-30. doi: 10.1111/j.1423-0410.2009.01273.x. PMID 20432513
- [Background] Masser B. Experienced donors, adverse events, and retention. Transfusion. 2012 Sep;52(9):1844-8. doi: 10.1111/j.1537-2995.2012.03829.x. No abstract available. PMID 22946968
- [Background] Sinclair KS, Campbell TS, Carey PM, Langevin E, Bowser B, France CR. An adapted postdonation motivational interview enhances blood donor retention. Transfusion. 2010 Aug;50(8):1778-86. doi: 10.1111/j.1537-2995.2010.02618.x. Epub 2010 Apr 23. PMID 20456674
- [Background] May M, Jordan J. The osmopressor response to water drinking. Am J Physiol Regul Integr Comp Physiol. 2011 Jan;300(1):R40-6. doi: 10.1152/ajpregu.00544.2010. Epub 2010 Nov 3. PMID 21048076
- [Background] Schroeder C, Bush VE, Norcliffe LJ, Luft FC, Tank J, Jordan J, Hainsworth R. Water drinking acutely improves orthostatic tolerance in healthy subjects. Circulation. 2002 Nov 26;106(22):2806-11. doi: 10.1161/01.cir.0000038921.64575.d0. PMID 12451007
- [Background] Endo Y, Yamauchi K, Tsutsui Y, Ishihara Z, Yamazaki F, Sagawa S, Shiraki K. Changes in blood pressure and muscle sympathetic nerve activity during water drinking in humans. Jpn J Physiol. 2002 Oct;52(5):421-7. doi: 10.2170/jjphysiol.52.421. PMID 12533246
- [Background] Mathias CJ, Young TM. Water drinking in the management of orthostatic intolerance due to orthostatic hypotension, vasovagal syncope and the postural tachycardia syndrome. Eur J Neurol. 2004 Sep;11(9):613-9. doi: 10.1111/j.1468-1331.2004.00840.x. PMID 15379740
- [Background] Moreno IL, Pastre CM, Ferreira C, de Abreu LC, Valenti VE, Vanderlei LC. Effects of an isotonic beverage on autonomic regulation during and after exercise. J Int Soc Sports Nutr. 2013 Jan 4;10(1):2. doi: 10.1186/1550-2783-10-2. PMID 23286515
- [Background] Charkoudian N, Eisenach JH, Joyner MJ, Roberts SK, Wick DE. Interactions of plasma osmolality with arterial and central venous pressures in control of sympathetic activity and heart rate in humans. Am J Physiol Heart Circ Physiol. 2005 Dec;289(6):H2456-60. doi: 10.1152/ajpheart.00601.2005. Epub 2005 Sep 30. PMID 16199481
- [Background] Ditto B, France CR, Albert M, Byrne N. Dismantling applied tension: mechanisms of a treatment to reduce blood donation-related symptoms. Transfusion. 2007 Dec;47(12):2217-22. doi: 10.1111/j.1537-2995.2007.01449.x. Epub 2007 Aug 21. PMID 17714419